CLINICAL TRIAL: NCT04079231
Title: A Comparative Double Masked, Two-Arm, Randomized, Multicenter, Phase IIIb Study Analyzing the Efficacy and Safety of Brolucizumab Versus Aflibercept in Patients With Visual Impairment Due to Diabetic Macular Edema (BUZZARD)
Brief Title: Efficacy and Safety of Brolucizumab vs. Aflibercept in Patients With Visual Impairment Due to Diabetic Macular Edema
Acronym: BUZZARD
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: This study was cancelled due to COVID-19.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRTH258BDE01
Record Dates: First submitted 2019-08-12; First posted 2019-09-06 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-01

CONDITIONS: Diabetic Macula Edema
Keywords: Diabetic Macula Edema; Intravitreal injection; brolucizumab; aflibercept; double-masked
MeSH Terms: interventions — brolucizumab; aflibercept

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brolucizumab 6 mg (Experimental): Brolucizumab 6 mg/0.05 mL, 5 loading doses, with subsequent doses per protocol-specified maintenance schedule
  Interventions: Drug: Brolucizumab
- Aflibercept 2 mg (Active Comparator): Aflibercept 2 mg/0.05 mL, as labeled, 5 loading doses, with subsequent doses every 8 weeks
  Interventions: Drug: Aflibercept

INTERVENTIONS:
Drug: Brolucizumab — Intravitreal Injection
  Other Names: RTH258, ESBA1008
  Arms: Brolucizumab 6 mg
Drug: Aflibercept — Intravitreal injection
  Other Names: Eylea
  Arms: Aflibercept 2 mg

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of brolucizumab in treatment of patients with visual impairment due to diabetic macular edema (DME).

DETAILED DESCRIPTION:
In this 48-week, randomized, double-masked, multicenter, active controlled study, consenting patients will be randomized in a 1:1 ratio to one of the two treatment arms and attend 14 planned visits.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 or type 2 diabetes mellitus and HbA1c of ≤10% at Screening
* BCVA score between 23 and 65 letters, inclusive, using ETDRS visual acuity testing charts at a testing distance of 4 meters (approximate Snellen equivalent of 20/50 to 20/320), at screening and baseline
* DME involving the center of the macula, with central subfield retinal thickness (measured from RPE to ILM inclusively) of ≥ 320 µm on SD-OCT

Exclusion Criteria:

* High risk or advanced proliferative diabetic retinopathy in the study eye as per reading Center
* Active intraocular or periocular infection or active intraocular inflammation in the study eye
* Uncontrolled glaucoma in the study eye defined as intraocular pressure (IOP) > 25 millimeters mercury (mmHg)
* Previous treatment with any anti-VEGF drugs or investigational drugs in the study eye in the last 3 months prior randomization
* Stroke or myocardial infarction during the 6-month period prior to baseline
* Uncontrolled blood pressure defined as a systolic value ≥160 mmHg or diastolic value ≥100 mmHg Other protocol-specified inclusion/exclusion criteria may apply

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a gain in Best Corrected Visual Acurity (BCVA) of ≥15 ETDRS letters at week 48 | Week 48
  BCVA will be assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts
Mean change in BCVA from baseline to Week 48 | Baseline, Week 48
  BCVA will be assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts

SECONDARY OUTCOMES:
Change from baseline in BCVA averaged over a period Week 36 to Week 48 | Week 36, Week 48
  BCVA will be assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts
Proportion of patients with a gain in BCVA of ≥10 ETDRS letters from baseline to Week 48 | Baseline, Week 48
  BCVA will be assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts
Proportion of patients with a loss in BCVA of ≥15 ETDRS letters from baseline to Week 48 | Baseline, Week 48
  BCVA will be assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts
Proportion of patients with a loss in BCVA of ≥10 ETDRS letters from baseline to Week 48 | Baseline, Week 48
  BCVA will be assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts
Proportion of patients maintained at q12w up to Week 48 | Baseline, Week 48
  Percentage of participants maintained at q12w (quarterly, every 12 weeks). This outcome measure is pre-specified for brolucizumab treatment arm only
Proportion of patients maintained at q12w up to Week 48, within those patients that qualified for q12w at week 28 | Week 28, Week 48
  Percentage of patients maintained at (q12w) quarterly, every 12 weeks, up to Week 48, within those patients that qualified for (q12w) at week 28. This outcome measure is pre-specified for brolucizumab treatment arm only
Change from baseline in central subfield thickness (CSFT, as determined by SD-OCT) at each assessment visit | Baseline, Week 48
  Assessed by Spectral Domain Optical Coherence Tomography (SD-OCT)
Average change in CSFT from baseline over the period Week 36 through Week 48 | Week 36, Week 48
  Assessed by Spectral Domain Optical Coherence Tomography (SD-OCT)
Average change in CSFT from baseline over the period Week 4 to Week 48 | Week 4, Week 48
  Assessed by Spectral Domain Optical Coherence Tomography (SD-OCT)
Patient status regarding normal CSFT thickness (<280 microns) at each assessment visit | Baseline, Week 48
  Assessed by Spectral Domain Optical Coherence Tomography (SD-OCT)
Change from baseline in Central Subfield Thickness-neurosensory (CSFTns, as determined by SD-OCT) at each assessment visit | Baseline, week 48
  Assessed by Spectral Domain Optical Coherence Tomography (SD-OCT)
Average change in CSFTns from baseline over the period Week 36 through Week 48 | Baseline, Week 36, Week 48
  Assessed by Spectral Domain Optical Coherence Tomography (SD-OCT)
Average change in CSFTns from baseline over the period Week 4 to Week 48 | Baseline, Week 4, Week 48
  Assessed by Spectral Domain Optical Coherence Tomography (SD-OCT)
Proportion of patients with presence of SRF, IRF and simultaneous absence of SRF and IRF at each assessment visit | Baseline, Week 48
  Assessed by Spectral Domain Optical Coherence Tomography (SD-OCT)
Proportion of patients with presence of leakage on FA at Week 48 | Week 48
  Assessed by fluorescein angiography
Change in ETDRS Diabetic Retinopathy Severity Scale (DRSS) score up to Week 48 (central reading) | Baseline, Week 48
  The Diabetic Retinopathy Disease Severity Scale measures the 5 levels of diabetic retinopathy - none, mild, moderate, severe, and proliferative
Patient status regarding a ≥2- and ≥3-step improvement or worsening from baseline in the ETDRS Diabetic Retinopathy Severity Scale (DRSS) score at each assessment visit | Baseline, Week 48
  Disease status measured by ETDRS-DRSS. Diabetic Retinopathy Severity Scale (DRSS) score at each assessment visit.
Incidence of progression to PDR as assessed by ETDRS-DRSS score of at least 61 by Week 48 | Baseline, Week 48
  Incidence of progression to proliferative diabetic retinopathy (PDR) measured by ETDRS-DRSS. Diabetic Retinopathy Severity Scale (DRSS) score at each assessment visit.
Rate of "inactive" PDRs by Week 48 compared to baseline | Baseline, Week 48
  Rate of "inactive" proliferative diabetic retinopathy (PDRs) by Week 48 compared to baseline as measured by Diabetic Retinopathy Severity Scale (DRSS) score.

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on ww.clinicalstudydatarequest.com.